CLINICAL TRIAL: NCT04926506
Title: Efficacy and Safety of Intramuscular Injection of Xiyanping Injection in the Treatment of Acute Bronchitis in Children: a Multicenter, Randomized, Parallel Controlled Clinical Study
Brief Title: Efficacy and Safety of Intramuscular Injection of Xiyanping Injection in the Treatment of Acute Bronchitis in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QF-XYP2021-1
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-06

CONDITIONS: Acute Bronchitis in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xiyanping injection combined with routine treatment (Experimental)
  Interventions: Drug: Xiyanping injection
- routine treatment (No Intervention)

INTERVENTIONS:
Drug: Xiyanping injection — Intramuscular injection of Xiyanping injection, 0.3mL / (kg.d) daily, Bid
  Arms: Xiyanping injection combined with routine treatment

SUMMARY:
Any pathogen that causes an upper respiratory tract infection can cause bronchitis.The primary pathogen is virus. On the basis of virus infection, pathogenic bacteria may cause secondary infection or co-infection。Xiyanping injection is mainly used in the treatment of bronchitis by intravenous injection。

DETAILED DESCRIPTION:
To further verify the clinical value and safety of intramuscular injection of Xiyanping injection in the treatment of acute bronchitis in children, provide reference for subsequent validation studies, and provide more reasonable and standard application guidance and basis for clinical practice.A multicenter, randomized, parallel controlled study was conducted on the treatment of acute bronchitis by intramuscular injection of Xiyanping injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1-6 years (>1 years, ≤6years);
2. Children who meet the diagnosis criteria of acute bronchitis in children;
3. All symptoms, including cough, had been present for less than 72 hours at the time of inclusion screening;
4. The informed consent process complies with the regulations, and the legal guardian signs the informed consent.

Exclusion Criteria:

1. Have used Chinese medicine injection containing andrographolide and similar functions (clearing heat and detoxifying, relieving cough and stopping dysentery) or oral dosage within 72 hours.
2. Children with severe bronchitis or early pneumonia;
3. Children with acute infectious diseases such as measles, pertussis,influenza and hand-foot-and-mouth disease;
4. Children with diseases such as acute upper respiratory tract infection, suppurative tonsillitis, wheezing bronchitis, bronchial asthma, bronchiolitis pneumonia, tuberculosis, tumor;
5. neutrophil granulocyte>80%, or those who need antibiotic therapy;
6. Children with severe malnutrition and immunodeficiency;
7. Children with severe primary diseases such as heart, liver, kidney, digestion and hematopoietic system;
8. Allergic constitution and children allergic to the drug used in this study;
9. Children who are taking epinephrine, isoproterenol and other catecholamines;
10. Children who are taking MAO inhibitors or tricyclic antidepressants
11. Children who are taking non-selective β-blockers such as Propranolol;
12. Those who are not included based on the investigators judgment.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-10-08 (Estimated); Primary Completion 2022-09-21 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Total clinical effective rate | up to day 7
  The children were evaluated according to the improvement of body temperature (axillary temperature), cough, expectoration, lung rales and other symptoms and signs and the improvement time

SECONDARY OUTCOMES:
Cough easing | up to day 7
  Symptoms are less than or equal to 1 point (mild) and remain for 24 hours or more
Lung rales relieved | up to day 7
  Symptoms are less than or equal to 1 point (mild) and remain for 24 hours or more
Fever relief | up to day 7
  Body temperature <37.5℃ (axillary temperature) and maintained for 24h or more